CLINICAL TRIAL: NCT07368309
Title: Clinical Management Strategies for Patients With Cirrhosis and Esophagogastric Varices Complicated by Early-stage Upper Gastrointestinal Cancer: a Multicenter Retrospective Cohort Study
Brief Title: Clinical Management Strategies for Patients With Cirrhosis and Esophagogastric Varices Complicated by Early-stage Upper Gastrointestinal Cancer
Status: Completed | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Southwest Hospital, China (Other); Shanxi Coal Central Hospital (Unknown); Beijing Friendship Hospital (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); Tongji Hospital Affiliated to Tongji Medical College of HUST (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, ChenMingkai, Department of Gastroenterology, Renmin Hospital of Wuhan University
Other Study IDs: WDRY2023-K116
Record Dates: First submitted 2026-01-11; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2024-12

CONDITIONS: Cirrhosis; Esophagogastric Varices; Early-stage Upper Gastrointestinal Cancer
Keywords: Cirrhosis; Endoscopic submucosal dissection; Esophagogastric varices; Early-stage upper gastrointestinal cancer
MeSH Terms: conditions — Fibrosis; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cirrhosis group: cirrhotic patients with EGV and early-stage upper gastrointestinal cancer 问who underwent ESD
- noncirrhosis group: Patients who underwent ESD without cirrhosis and EGV

SUMMARY:
Managing early-stage upper gastrointestinal cancer in patients with liver cirrhosis and esophagogastric varices (EGV) poses substantial clinical challenges. Although endoscopic submucosal dissection (ESD) is an established treatment for these early cancers, its efficacy and safety in this high-risk population are poorly defined. Therefore, this study aims to investigate optimal screening and treatment strategies for early-stage upper gastrointestinal cancer in cirrhotic patients with EGV. Perioperative outcomes were compared between the two groups.

DETAILED DESCRIPTION:
Oesophageal and gastric cancers remain leading causes of cancer-related morbidity and mortality worldwide. Early endoscopic screening is crucial, as it significantly improves prognosis. ESD has become the standard minimally invasive treatment for early-stage lesions because it enables en-bloc resection with rapid recovery and favourable cost-effectiveness.

In patients with liver cirrhosis and EGV, however, the management of early-stage upper gastrointestinal cancer is uniquely challenging. First, The detection of early-stage cancer depends on identifying subtle alterations in mucosal coloration and morphology, yet in cirrhotic patients these signs are masked by co-existing varices, portal-hypertensive gastropathy and accompanying mucosal changes, imposcope passage, obscuring inspection and raising the likelihood of missed cancers. Second, underlying coagulopathy and thrombocytopenia in these patients theoretically elevate the risk of procedure-related bleeding, especially when varices are adjacent to or located at the resection area. Presently, clinical guidelines provide no specific guidance for this high-risk population. Existing evidence is limited, derived mostly from small, single-arm studies. To establish a safe and effective standardized management protocol and to evaluate the feasibility of ESD in this setting, we conducted this multicentre, retrospective cohort study to inform clinical decision-making. This study was conducted at 7 tertiary hospitals in China. Consecutive patients who underwent ESD for early-stage upper gastrointestinal cancer between January 2018 and April 2023 were enrolled. Patients were stratified into a cirrhosis group (study group) and a noncirrhosis control group. Inclusion criteria for the study group were: age >18 years; a clinical diagnosis of liver cirrhosis; and endoscopically confirmed EGV. The noncirrhosis group comprised patients over 18 years with early-stage upper gastrointestinal cancer but without cirrhosis, randomly selected from the same pool. Common exclusion criteria were: concomitant end-stage disease of major organs (e.g., active malignancy, heart failure, respiratory failure) or an American Society of Anesthesiologists (ASA) physical status classification ≥ III; previous surgery for cirrhosis, EGV, or other upper gastrointestinal lesions; incomplete clinical records. Preoperative characteristics, demographic data, and perioperative management were compared between groups to inform the development of perioperative strategies for patients with cirrhosis and EGV. Trained investigators extracted demographic, laboratory, perioperative and postoperative outcome data from electronic medical records. Safety indicators included intra/postoperative adverse events, mortality, and ICU transfer. Efficacy indicators were en bloc resection rate, R0 resection rate, procedure time, and resection efficiency.

ELIGIBILITY:
Inclusion Criteria:

The cirrhosis group:

* Age >18 years;
* A clinical diagnosis of liver cirrhosis
* Endoscopically confirmed EGV.

The noncirrhosis group:

* Age > 18 years
* With early-stage upper gastrointestinal cancer but without cirrhosis

Exclusion Criteria:

* Concomitant end-stage disease of major organs (e.g., active malignancy, heart failure, respiratory failure) or an American Society of Anesthesiologists (ASA) physical status classification ≥ III
* Previous surgery for cirrhosis, EGV, or other upper gastrointestinal lesions
* Incomplete clinical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who underwent ESD for early-stage upper gastrointestinal cancer between January 2018 and April 2023 were enrolled. See the previous entry for specific eligibility criteria
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Mortality | Perioperative
  Patients who died due to ESD
ICU transfer | Perioperative
  Transferred to ICU due to ESD
Intraoperative major bleeding | Perioperative
  Intraoperative major bleeding was defined as active bleeding requiring specific endoscopic hemostasis
en bloc resection rate | Perioperative
  En bloc resection was complete removal of the lesion in one piece without fragmentation
R0 resection | Perioperative
  R0 resection was histopathological confirmation of tumour-free lateral and vertical margins
Delayed bleeding | Perioperative
  Delayed bleeding was defined as any evidence of gastrointestinal hemorrhage

SECONDARY OUTCOMES:
Other intra/postoperative adverse events | Perioperative
  Intraoperative perforation, fever, esophageal stricture, delayed perforation, pain, and nausea/vomiting
Procedure time | Perioperative
  ESD operation time
ESD efficiency | Perioperative
  The average time required to resect lesions per square centimeter

OTHER OUTCOMES:
Other cirrhosis complication | Perioperative
  New complications of liver cirrhosis due to ESD surgery
Hospitalization duration | Perioperative
  The duration of hospitalization due to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Chen, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
The patients included in the study are rare, and the data are precious and difficult to collect. However, if any researcher needs our data for secondary analysis (systematic review, etc.) after publication, they can contact us by email.